CLINICAL TRIAL: NCT05918822
Title: A Phase 1, Open-Label, Randomized, Two-Part Study in Healthy Adult Participants to Evaluate the Relative Bioavailability of Maribavir Pediatric Formulation Compared to the Commercial Formulation, as Well as, Food Effect, and Rabeprazole Gastric Acid-Reducing Effect on the Pharmacokinetics of Single-Dose Maribavir Pediatric Formulation
Brief Title: A Study of Maribavir Pediatric Formulation in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TAK-620-1024
Record Dates: First submitted 2023-06-16; First posted 2023-06-26 (Actual); Results first posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-06

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Rabeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (8):
- Part 1, Sequence 1: Treatment A + Treatment B + Treatment C (Experimental): Participants will receive maribavir single 200 mg commercial tablet, on Day 1 of Treatment Period 1 under fasting condition (Treatment A), followed by maribavir 200 mg pediatric powder-for-oral suspension, single oral dose on Day 1 of Treatment Period 2 under fasting condition (Treatment B), and further followed by maribavir 200 mg pediatric powder-for-oral suspension, single oral dose on Day 1 of Treatment Period 3 administered with a high fat/high calorie meal (Treatment C). There will be a washout period of a minimum of 72 hours between each treatment.
  Interventions: Drug: Maribavir Commercial Tablet Formulation; Drug: Maribavir Pediatric Powder-for-oral Suspension Formulation
- Part 1, Sequence 2: Treatment A + Treatment C + Treatment B (Experimental): Participants will receive maribavir single 200 mg commercial tablet, on Day 1 of Treatment Period 1 under fasting condition (Treatment A), followed by maribavir 200 mg pediatric powder-for-oral suspension, single oral dose on Day 1 of Treatment Period 2 administered with a high fat/high calorie meal (Treatment C), and further followed by maribavir 200 mg pediatric powder-for-oral suspension, single oral dose on Day 1 of Treatment Period 3 under fasting condition (Treatment B). There will be a washout period of a minimum of 72 hours between each treatment.
  Interventions: Drug: Maribavir Commercial Tablet Formulation; Drug: Maribavir Pediatric Powder-for-oral Suspension Formulation
- Part 1, Sequence 3: Treatment B + Treatment A + Treatment C (Experimental): Participants will receive maribavir 200 mg pediatric powder-for-oral suspension, single oral dose on Day 1 of Treatment Period 1 under fasting condition (Treatment B), followed by maribavir single 200 mg commercial tablet, on Day 1 of Treatment Period 2 under fasting condition (Treatment A), and further followed by maribavir 200 mg pediatric powder-for-oral suspension, single oral dose on Day 1 of Treatment Period 3 administered with a high fat/high calorie meal (Treatment C). There will be a washout period of a minimum of 72 hours between each treatment.
  Interventions: Drug: Maribavir Commercial Tablet Formulation; Drug: Maribavir Pediatric Powder-for-oral Suspension Formulation
- Part 1, Sequence 4: Treatment B + Treatment C + Treatment A (Experimental): Participants will receive maribavir 200 mg pediatric powder-for-oral suspension, single oral dose on Day 1 of Treatment Period 1 under fasting condition (Treatment B), followed by maribavir 200 mg pediatric powder-for-oral suspension, single oral dose on Day 1 of Treatment Period 2 administered with a high fat/high calorie meal (Treatment C), and further followed by maribavir single 200 mg commercial tablet, on Day 1 of Treatment Period 3 under fasting condition (Treatment A). There will be a washout period of a minimum of 72 hours between each treatment.
  Interventions: Drug: Maribavir Commercial Tablet Formulation; Drug: Maribavir Pediatric Powder-for-oral Suspension Formulation
- Part 1, Sequence 5: Treatment C + Treatment A + Treatment B (Experimental): Participants will receive maribavir 200 mg pediatric powder-for-oral suspension, single oral dose on Day 1 of Treatment Period 1 administered with a high fat/high calorie meal (Treatment C), followed by maribavir single 200 mg commercial tablet, on Day 1 of Treatment Period 2 under fasting condition (Treatment A), and further followed by maribavir 200 mg pediatric powder-for-oral suspension, single oral dose on Day 1 of Treatment Period 3 under fasting condition (Treatment B). There will be a washout period of a minimum of 72 hours between each treatment.
  Interventions: Drug: Maribavir Commercial Tablet Formulation; Drug: Maribavir Pediatric Powder-for-oral Suspension Formulation
- Part 1, Sequence 6: Treatment C + Treatment B+ Treatment A (Experimental): Participants will receive maribavir 200 mg pediatric powder-for-oral suspension, single oral dose on Day 1 of Treatment Period 1 administered with a high fat/high calorie meal (Treatment C), followed by maribavir 200 mg pediatric powder-for-oral suspension, single oral dose on Day 1 of Treatment Period 2 under fasting condition (Treatment B), and further followed by maribavir single 200 mg commercial tablet, on Day 1 of Treatment Period 3 under fasting condition as (Treatment A). There will be a washout period of a minimum of 72 hours between each treatment.
  Interventions: Drug: Maribavir Commercial Tablet Formulation; Drug: Maribavir Pediatric Powder-for-oral Suspension Formulation
- Part 2: Treatment D: maribavir 200 mg (Experimental): Participants will receive maribavir 200 mg pediatric powder-for-oral suspension, single oral dose on Day 1 of Treatment Period 1 under fasting condition (Treatment D).
  Interventions: Drug: Maribavir Pediatric Powder-for-oral Suspension Formulation
- Part 2, Treatment E: rabeprazole 20 mg + maribavir 200 mg (Experimental): Participants will receive rabeprazole single 20 mg tablet, once daily on Days 1 to 5 of Treatment Period 2 under fasting condition followed by maribavir 200 mg pediatric powder-for-oral suspension, single oral dose, 2 hours after rabeprazole dosing on morning of Day 5 of Treatment Period 2 under fasting condition (Treatment E). There will be a washout period of a minimum of 72 hours between maribavir dosing in Treatment Period 1 and first dose of rabeprazole in Treatment Period 2.
  Interventions: Drug: Maribavir Pediatric Powder-for-oral Suspension Formulation; Drug: Rabeprazole

INTERVENTIONS:
Drug: Maribavir Commercial Tablet Formulation — Maribavir commercial tablet.
  Other Names: TAK-620
  Arms: Part 1, Sequence 1: Treatment A + Treatment B + Treatment C; Part 1, Sequence 2: Treatment A + Treatment C + Treatment B; Part 1, Sequence 3: Treatment B + Treatment A + Treatment C; Part 1, Sequence 4: Treatment B + Treatment C + Treatment A; Part 1, Sequence 5: Treatment C + Treatment A + Treatment B; Part 1, Sequence 6: Treatment C + Treatment B+ Treatment A
Drug: Maribavir Pediatric Powder-for-oral Suspension Formulation — Maribavir pediatric powder-for-oral suspension.
  Other Names: TAK-620
Drug: Rabeprazole — Rabeprazole tablet.
  Arms: Part 2, Treatment E: rabeprazole 20 mg + maribavir 200 mg

SUMMARY:
The study will have 2 parts, Part 1 and Part 2. Participants will only participate in one part.

The main aim of Part 1 of this study is to check the ability of a single dose of maribavir pediatric formulation to be absorbed in the digestive tract compared to commercial tablet formulation and to check how a high-fat, high-calorie meal affects absorption, distribution, and elimination of maribavir pediatric formulation given orally as water suspension.

The main aim of Part 2 of this study is to assess the stomach acid reducing effect of multiple doses of rabeprazole on absorption, distribution, and elimination of maribavir pediatric formulation given orally as water suspension.

Each participant will stay in the study clinic from the day before the first treatment until the day after the last treatment.

DETAILED DESCRIPTION:
Part 1 is a crossover design with three treatments (Treatments A, B, and C), six sequences, and three periods.

The relative bioavailability of 200 milligrams (mg) maribavir pediatric formulation administered orally as water suspension under fasting conditions (Treatment B) will be compared to 200 mg maribavir commercial tablet administered orally under fasting conditions (Treatment A). In addition, the effect of food on the pharmacokinetics (PK) of 200 mg maribavir pediatric formulation administered orally as water suspension under fasting conditions (Treatment B) and fed conditions (Treatment C) will be assessed. In each sequence, participants will receive three treatments (Treatments A, B, and C) per schedule.

* Sequence 1: Treatment A + Treatment B + Treatment C
* Sequence 2: Treatment A + Treatment C + Treatment B
* Sequence 3: Treatment B + Treatment A + Treatment C
* Sequence 4: Treatment B + Treatment C + Treatment A
* Sequence 5: Treatment C + Treatment A + Treatment B
* Sequence 6: Treatment C + Treatment B + Treatment A

Part 2 is a single fixed-sequence design with two treatments (Treatments D and E). The two treatments will be administered to evaluate the gastric acid-reducing effect of multiple doses of rabeprazole on the PK of a single dose of 200 mg maribavir pediatric formulation administered orally as water suspension.

ELIGIBILITY:
Inclusion Criteria:

* An understanding, ability, and willingness to fully comply with study procedures and restrictions and to voluntarily sign (personally or via a legally authorized representative) informed consent form to participate in the study.
* Age 18 to 55 years, inclusive at the time of consent, at the screening visit.
* Male, or non-pregnant, non-breastfeeding female who agrees to comply with any applicable contraceptive requirements of the protocol or female of non-childbearing potential.
* Body mass index (BMI) between 18.0 and 30.0 kilogram per meter square (kg/m^2), inclusive with a body weight greater than (>) 50 kilograms (kg) (110 pounds [lbs]), at the screening visit.
* Healthy as determined by the Investigator or designee on the basis of screening evaluations and medical history.
* Hemoglobin for males greater than or equal to (>=) 135.0 gram per liter (g/L) and females >=120.0 g/L, at the screening visit and on Day -1 of Treatment Period 1.
* Ability to swallow a dose of maribavir or rabeprazole.

Exclusion Criteria:

* History or presence of gastritis, gastrointestinal (GI) tract disorder, hepatic disorder or cholecystectomy, history of treated or untreated Helicobacter pylori, ulcer disease or other clinical condition which, in the opinion of the investigator or designee, may affect the absorption, distribution, metabolism, or elimination of the study drugs.
* History of any hematological, hepatic, respiratory, cardiovascular, renal, neurological or psychiatric disease, gall bladder removal, or current recurrent disease that could affect the action, absorption, or disposition of the study drugs, or clinical or laboratory assessments.
* Current or relevant history of physical or psychiatric illness, any medical disorder that may require treatment or make the participant unlikely to fully complete the study, or any condition that presents undue risk from the study drugs or procedures.
* Known or suspected intolerance or hypersensitivity to maribavir or rabeprazole (Part 2 only), closely related compounds, or any of the stated ingredients and excipients.
* Significant illness, as judged by the Investigator or designee, within 2 weeks of the first dose of the investigational drug (ID).
* Has diarrhea within 4 hours of the first dose of the ID.
* Donation of blood or blood products (example, plasma or platelets) within 60 days prior to receiving the first dose of the ID.
* Within 30 days prior to the first dose of the ID:

  * Have used any investigational product (if elimination half-life is less than [<] 6 days, otherwise 5 half-lives).
  * Have been enrolled in a clinical study (including vaccine studies) that, in the Investigator or designee's opinion, may impact this Takeda-sponsored study.
  * Have had any substantial changes in eating habits, as assessed by the Investigator or designee.
* Systolic blood pressure >140 millimeters of mercury (mmHg) or <90 mmHg, and/or diastolic blood pressure >90 mmHg or <50 mmHg, at the screening visit.
* Corrected QT interval (QTc) >450 millisecond (msec) at the screening visit. If QTc exceeds 450 msec, the ECG should be repeated two more times and the average of the three QTc values should be used to determine the participant's eligibility.
* Known history of alcohol or other substance abuse within the last year.
* Male participants who consume more than 21 units of alcohol per week or three units per day. Female participants who consume more than 14 units of alcohol per week or two units per day (one alcohol unit = one beer or one wine [5 ounces [oz]/150 milliliter [mL]] or one liquor [1.5 oz/40 mL] or 0.75 oz alcohol).
* A positive screen for alcohol or drugs of abuse at the screening visit or on Day -1 of Treatment Period 1. Urine samples are to be tested for amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, methadone, opiates, and phencyclidine.
* A positive Human immunodeficiency virus (HIV), Hepatitis B surface antigen (HBsAg), or Hepatitis C virus (HCV) antibody screen at the screening visit.
* Use of tobacco in any form (example, smoking or chewing) or other nicotine-containing products in any form (example, gum, patch). Ex-users must self-report that they have stopped using tobacco for at least 3 months prior to receiving the first dose.
* Routine consumption of more than two units of caffeine per day or participants who experience caffeine withdrawal headaches (One caffeine unit is contained in the following items: one 6-oz [180 mL] cup of coffee, two 12-oz [360 mL] cans of cola, one 12-oz cup of tea, three 1-oz [85 grams [g]] chocolate bars). Decaffeinated coffee, tea, or cola are not considered to contain caffeine.
* Current use of any prescription medication with the exception of hormonal contraceptives and hormonal replacement therapy. Current use of any over-the-counter (OTC) medication (including OTC multi-vitamin, herbal, or homeopathic preparations) within 14 days of the first dose. Hormonal contraceptives and hormonal replacement therapy may be permitted if the female participant has been on the same stable dose for at least 3 months prior to first dose.
* Current use of antacids, proton pump inhibitors (PPIs), or histamine type 2 (H2) antagonists within 14 days of the first dose, except for on-study rabeprazole.
* Inability or unwillingness to consume 100 percent of the high-fat, high-calorie meal (including participants with lactose or gluten intolerance).
* Female participants with a positive pregnancy test at the screening visit or on Day -1 of Treatment Period 1 or who are lactating.
* Participants on a diet incompatible with the on-study diet, in the opinion of the Investigator or designee, within the 30 days prior to the first dosing and throughout the study.
* Recent history (within 1 month) of oral/nasal cavity infections, history of gastroesophageal reflux, asthma treatment with albuterol, or zinc supplementation.
* Participants with dry mouth syndrome or burning mouth syndrome or participants suffering from dysgeusia.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2023-07-25 (Actual); Primary Completion 2023-08-25 (Actual); Study Completion 2023-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Celerion, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/837e7f476b7a4922??page=1&idFilter=TAK-620-1024

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at single center in the United States from 25 July 2023 to 01 September 2023.
Pre-assignment Details: A total of 32 participants were enrolled and randomized in this 2-part (18 in Part 1 and 14 in Part 2) study. Part 1 consisted of 3 treatment-periods and participants were randomized into one of 6 treatment sequences: ABC, ACB, BAC, BCA, CAB, or CBA. Part 2 consisted of 2-treatment periods and was a single fixed-sequence design with 2 treatments: Treatment D and E.
Groups:
- Part 1, Sequence 1: Treatment A + Treatment B + Treatment C: On Day 1 of Treatment Period 1, participants received maribavir single 200 milligrams (mg) commercial tablet, under fasting conditions (Treatment A). On Day 1 of Treatment Period 2, participants received single oral dose of maribavir 200 mg pediatric powder-for-oral suspension under fasting conditions (Treatment B). On Day 1 of Treatment Period 3, participants received single oral dose of maribavir 200 mg pediatric powder-for-oral suspension administered with a high fat/high calorie meal (Treatment C). There was a washout period of a minimum of 3 days between each Treatment Period.
- Part 1, Sequence 2: Treatment A + Treatment C + Treatment B: On Day 1 of Treatment Period 1, participants received maribavir single 200 mg commercial tablet under fasting conditions (Treatment A), followed by single oral dose of maribavir 200 mg pediatric powder-for-oral suspension on Day 1 of Treatment Period 2 administered with a high fat/high calorie meal (Treatment C), and further followed by single oral dose of maribavir 200 mg pediatric powder-for-oral suspension on Day 1 of Treatment Period 3 under fasting conditions (Treatment B). There was a washout period of a minimum of 3 days between each Treatment Period.
- Part 1, Sequence 3: Treatment B + Treatment A + Treatment C: On Day 1 of Treatment Period 1, participants received a single oral dose of maribavir 200 mg pediatric powder-for-oral suspension under fasting conditions (Treatment B). On Day 1 of Treatment Period 2, participants received maribavir single 200 mg commercial tablet under fasting conditions (Treatment A). On Day 1 of Treatment Period 3, participants received single oral dose of maribavir 200 mg pediatric powder-for-oral suspension administered with a high fat/high calorie meal (Treatment C). There was a washout period of a minimum of 3 days between each Treatment Period.
- Part 1, Sequence 4: Treatment B + Treatment C + Treatment A: On Day 1 of Treatment Period 1, participants received single oral dose of maribavir 200 mg pediatric powder-for-oral suspension under fasting conditions (Treatment B). On Day 1 of Treatment Period 2 participants received single oral dose of maribavir 200 mg pediatric powder-for-oral suspension administered with a high fat/high calorie meal (Treatment C). On Day 1 of Treatment Period 3, participants received maribavir single 200 mg commercial tablet under fasting conditions (Treatment A). There was a washout period of a minimum of 3 days between each Treatment Period.
- Part 1, Sequence 5: Treatment C + Treatment A + Treatment B: On Day 1 of Treatment Period 1, participants received maribavir 200 mg pediatric powder-for-oral suspension, single oral dose administered with a high fat/high calorie meal (Treatment C). On Day 1 of Treatment Period 2, participants received maribavir single 200 mg commercial tablet under fasting conditions (Treatment A). On Day 1 of Treatment Period 3, participants received single oral dose of maribavir 200 mg pediatric powder-for-oral suspension under fasting conditions (Treatment B). There was a washout period of a minimum of 3 days between each Treatment Period.
- Part 1, Sequence 6: Treatment C + Treatment B+ Treatment A: On Day 1 of Treatment Period 1, participants received maribavir 200 mg pediatric powder-for-oral suspension, single oral dose administered with a high fat/high calorie meal (Treatment C). On Day 1 of Treatment Period 2, participants received single oral dose of maribavir 200 mg pediatric powder-for-oral suspension under fasting conditions (Treatment B). On Day 1 of Treatment Period 3, participants received maribavir single 200 mg commercial tablet under fasting conditions (Treatment A). There was a washout period of a minimum of 3 days between each Treatment Period.
- Part 2: Treatment D + E: Maribavir 200 mg + Rabeprazole 20 mg: On Day 1 of Treatment Period 1, participants received a single oral dose of 200 mg maribavir powder-for-oral suspension formulation under fasting conditions (Treatment D). On Days 1 to 5 of Treatment Period 2, participants received oral doses of 20 mg rabeprazole, once daily, under fasting conditions. On the morning of Day 5 of Treatment Period 2, two hours after rabeprazole dosing, participants received a single oral dose of 200 mg maribavir powder-for-oral suspension formulation under fasting conditions (Treatment E). There was a washout period of a minimum of 3 days between maribavir dosing in Treatment Period 1 and first dose of rabeprazole in Treatment Period 2.
Period: Treatment Period 1 (Part 1 and 2: 1 Day)
Arm/Group | Part 1, Sequence 1: Treatment A + Treatment B + Treatment C | Part 1, Sequence 2: Treatment A + Treatment C + Treatment B | Part 1, Sequence 3: Treatment B + Treatment A + Treatment C | Part 1, Sequence 4: Treatment B + Treatment C + Treatment A | Part 1, Sequence 5: Treatment C + Treatment A + Treatment B | Part 1, Sequence 6: Treatment C + Treatment B+ Treatment A | Part 2: Treatment D + E: Maribavir 200 mg + Rabeprazole 20 mg
Started | 3 | 3 | 3 | 3 | 3 | 3 | 14
Completed | 3 | 3 | 3 | 3 | 3 | 3 | 14
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 1 (Part 1 and 2: 3 Days)
Arm/Group | Part 1, Sequence 1: Treatment A + Treatment B + Treatment C | Part 1, Sequence 2: Treatment A + Treatment C + Treatment B | Part 1, Sequence 3: Treatment B + Treatment A + Treatment C | Part 1, Sequence 4: Treatment B + Treatment C + Treatment A | Part 1, Sequence 5: Treatment C + Treatment A + Treatment B | Part 1, Sequence 6: Treatment C + Treatment B+ Treatment A | Part 2: Treatment D + E: Maribavir 200 mg + Rabeprazole 20 mg
Started | 3 | 3 | 3 | 3 | 3 | 3 | 14
Completed | 3 | 3 | 3 | 3 | 3 | 3 | 14
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period2Part1:1Day;Part2:Day1-5
Arm/Group | Part 1, Sequence 1: Treatment A + Treatment B + Treatment C | Part 1, Sequence 2: Treatment A + Treatment C + Treatment B | Part 1, Sequence 3: Treatment B + Treatment A + Treatment C | Part 1, Sequence 4: Treatment B + Treatment C + Treatment A | Part 1, Sequence 5: Treatment C + Treatment A + Treatment B | Part 1, Sequence 6: Treatment C + Treatment B+ Treatment A | Part 2: Treatment D + E: Maribavir 200 mg + Rabeprazole 20 mg
Started | 3 | 3 | 3 | 3 | 3 | 3 | 14
Completed | 3 | 3 | 3 | 3 | 3 | 3 | 14
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 2 (Part 1 Only: 3 Days)
Arm/Group | Part 1, Sequence 1: Treatment A + Treatment B + Treatment C | Part 1, Sequence 2: Treatment A + Treatment C + Treatment B | Part 1, Sequence 3: Treatment B + Treatment A + Treatment C | Part 1, Sequence 4: Treatment B + Treatment C + Treatment A | Part 1, Sequence 5: Treatment C + Treatment A + Treatment B | Part 1, Sequence 6: Treatment C + Treatment B+ Treatment A | Part 2: Treatment D + E: Maribavir 200 mg + Rabeprazole 20 mg
Started | 3 | 3 | 3 | 3 | 3 | 3 | 0
Completed | 3 | 3 | 3 | 3 | 3 | 3 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 3 (Part 1 Only: 1 Day)
Arm/Group | Part 1, Sequence 1: Treatment A + Treatment B + Treatment C | Part 1, Sequence 2: Treatment A + Treatment C + Treatment B | Part 1, Sequence 3: Treatment B + Treatment A + Treatment C | Part 1, Sequence 4: Treatment B + Treatment C + Treatment A | Part 1, Sequence 5: Treatment C + Treatment A + Treatment B | Part 1, Sequence 6: Treatment C + Treatment B+ Treatment A | Part 2: Treatment D + E: Maribavir 200 mg + Rabeprazole 20 mg
Started | 3 | 3 | 3 | 3 | 3 | 3 | 0
Completed | 3 | 3 | 3 | 3 | 3 | 3 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety set included all participants who received at least one dose of maribavir.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1, Sequence 1: Treatment A + Treatment B + Treatment C | Part 1, Sequence 2: Treatment A + Treatment C + Treatment B | Part 1, Sequence 3: Treatment B + Treatment A + Treatment C | Part 1, Sequence 4: Treatment B + Treatment C + Treatment A | Part 1, Sequence 5: Treatment C + Treatment A + Treatment B | Part 1, Sequence 6: Treatment C + Treatment B+ Treatment A | Part 2: Treatment D + E: Maribavir 200 mg + Rabeprazole 20 mg | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 14 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 3 | 3 | 3 | 3 | 14 | 32
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2 | 2 | 2 | 1 | 6 | 15
  Male | 2 | 2 | 1 | 1 | 1 | 2 | 8 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 2 | 1 | 3 | 2 | 9 | 21
  Not Hispanic or Latino | 0 | 2 | 1 | 2 | 0 | 1 | 5 | 11
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 1 | 0 | 0 | 0 | 4 | 8
  White | 2 | 1 | 1 | 3 | 3 | 3 | 10 | 23
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Parts 1 and 2: Maximum Observed Plasma Concentration (Cmax) of Maribavir
Description: Cmax was defined as maximum observed concentration of maribavir in plasma.
Time Frame: Part 1 Day 1 and Part 2 Treatment D Day 1 and Treatment E Day 5: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16 and 24 hours post-dose
Population: Pharmacokinetic (PK) set included all participants who received at least one dose of maribavir, did not vomit or had diarrhea within four hours of the maribavir dosing, and had five or more post-dose time points with evaluable post-dose maribavir concentration values that enabled non-compartmental analysis (NCA).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (mcg/mL)
Groups:
- Part 1, Treatment A: Maribavir 200 mg: On Day 1 of Treatment Period 1, 2 and 3, participants received maribavir single 200 mg commercial tablet under fasting conditions.
- Part 1, Treatment B: Maribavir 200 mg: On Day 1 of Treatment Period 1, 2 and 3, participants received single oral dose of maribavir 200 mg pediatric powder-for-oral suspension under fasting conditions.
- Part 1, Treatment C: Maribavir 200 mg: On Day 1 of Treatment Period 1, 2 and 3, participants received maribavir 200 mg pediatric powder-for-oral suspension administered with a high fat/high calorie meal.
- Part 2, Treatment D: Maribavir 200 mg: On Day 1 of Treatment Period 1, participants received maribavir 200 mg pediatric powder-for-oral suspension under fasting conditions.
- Part 2, Treatment E: Rabeprazole 20 mg + Maribavir 200 mg: On Days 1 to 5 of Treatment Period 2, participants received oral doses of 20 mg rabeprazole, once daily, under fasting conditions. On the morning of Day 5 of Treatment Period 2, two hours after rabeprazole dosing, participants received a single oral dose of 200 mg maribavir powder-for-oral suspension formulation under fasting conditions.
Arm/Group | Part 1, Treatment A: Maribavir 200 mg | Part 1, Treatment B: Maribavir 200 mg | Part 1, Treatment C: Maribavir 200 mg | Part 2, Treatment D: Maribavir 200 mg | Part 2, Treatment E: Rabeprazole 20 mg + Maribavir 200 mg
Number analyzed (Participants) | 18 | 18 | 18 | 14 | 14
microgram per milliliter (mcg/mL) | 12.6 (26.3) | 10.4 (26.2) | 5.98 (28.3) | 10.2 (19.9) | 4.98 (49.9)
Statistical Analysis 1: Comparison: Part 1, Treatment A: Maribavir 200 mg vs Part 1, Treatment B: Maribavir 200 mg; Comparison of Cmax of Maribavir: Part 1: Treatment B (Test) versus Treatment A (Reference); Test type: Other — A mixed-effects model was applied to log (ln)-transformed plasma maribavir Cmax with treatment, period, and sequence as fixed effects, and participant within sequence as random effect. Point estimates and their associated 90% confidence intervals (CIs) were constructed for differences between Treatment B (test) versus Treatment A (reference). Point estimate and their associated 90% CIs were then back transformed to provide point estimates and 90% CIs for ratios of Treatment B versus Treatment A; Geometric Mean Ratio (GMR) (%) = 82.19, 90% CI 2-sided [74.31 to 90.91] — GMR (%) was calculated as 100*(Test/Reference)
Statistical Analysis 2: Comparison: Part 1, Treatment B: Maribavir 200 mg vs Part 1, Treatment C: Maribavir 200 mg; Comparison of Cmax of Maribavir: Part 1: Treatment C (Test) versus Treatment B (Reference); Test type: Other — A mixed-effects model was applied to ln-transformed plasma maribavir Cmax with treatment, period, and sequence as fixed effects, and participant within sequence as a random effect. Point estimates and their associated 90 percent (%) CIs were constructed for differences between Treatment C (test) versus Treatment B (reference). Point estimates and their associated 90% CIs were then back transformed to provide point estimates and 90% CIs for ratios of Treatment C versus Treatment B; Geometric Mean Ratio (GMR) (%) = 57.72, 90% CI 2-sided [52.18 to 63.84] — GMR (%) was calculated as 100*(Test/Reference)
Statistical Analysis 3: Comparison: Part 2, Treatment D: Maribavir 200 mg vs Part 2, Treatment E: Rabeprazole 20 mg + Maribavir 200 mg; Comparison of Cmax of Maribavir: Part 2: Treatment E (Test) versus Treatment D (Reference); Test type: Other — A mixed-effects model was applied to ln-transformed plasma maribavir Cmax with treatment as a fixed effect, and participant as a random effect. Point estimates and their associated 90% CIs were constructed for the differences between Treatment E (test) versus Treatment D (reference). The point estimates and their associated 90% CIs were then back transformed to provide point estimates and 90% CIs for the ratios of Treatment E versus Treatment D; Geometric Mean Ratio (GMR) (%) = 49.03, 90% CI 2-sided [40.07 to 60.00] — GMR (%) was calculated as 100*(Test/Reference)

2. Primary Outcome: Parts 1 and 2: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration (AUClast) of Maribavir
Description: AUClast was defined as the area under the concentration-time curve from time 0 to the time of the last quantifiable concentration of maribavir in plasma.
Time Frame: as for outcome 1
Population: PK set included all participants who received at least one dose of maribavir, did not vomit or had diarrhea within four hours of the maribavir dosing, and had five or more post-dose time points with evaluable post-dose maribavir concentration values that enabled NCA.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*hour per milliliter (mcg*h/mL)
Arm/Group | Part 1, Treatment A: Maribavir 200 mg | Part 1, Treatment B: Maribavir 200 mg | Part 1, Treatment C: Maribavir 200 mg | Part 2, Treatment D: Maribavir 200 mg | Part 2, Treatment E: Rabeprazole 20 mg + Maribavir 200 mg
Number analyzed (Participants) | 18 | 18 | 18 | 14 | 14
microgram*hour per milliliter (mcg*h/mL) | 55.5 (52.6) | 54.2 (50.2) | 44.4 (51.9) | 53.9 (37.3) | 37.7 (36.8)
Statistical Analysis 1: Comparison: Part 1, Treatment A: Maribavir 200 mg vs Part 1, Treatment B: Maribavir 200 mg; Comparison of AUClast of Maribavir: Part 1: Treatment B (Test) versus Treatment A (Reference); Test type: Other — A mixed-effects model was applied to ln-transformed plasma maribavir AUClast with treatment, period, and sequence as fixed effects, and participant within sequence as a random effect. Point estimates and their associated 90% CIs were constructed for differences between Treatment B (test) versus Treatment A (reference). Point estimates and their associated 90% CIs were then back transformed to provide point estimates and 90% CIs for ratios of Treatment B versus Treatment A; Geometric Mean Ratio (GMR) (%) = 97.59, 90% CI 2-sided [91.39 to 104.20] — GMR (%) was calculated as 100*(Test/Reference)
Statistical Analysis 2: Comparison: Part 1, Treatment B: Maribavir 200 mg vs Part 1, Treatment C: Maribavir 200 mg; Comparison of AUClast of Maribavir: Part 1: Treatment C (Test) versus Treatment B (Reference); Test type: Other — A mixed-effects model was applied to ln-transformed plasma maribavir AUClast with treatment, period, and sequence as fixed effects, and participant within sequence as a random effect. Point estimates and their associated 90% CIs were constructed for differences between Treatment C (test) versus Treatment B (reference). Point estimates and their associated 90% CIs were then back transformed to provide point estimates and 90% CIs for ratios of Treatment C versus Treatment B; Geometric Mean Ratio (GMR) (%) = 82.05, 90% CI 2-sided [76.84 to 87.61] — GMR (%) was calculated as 100*(Test/Reference)
Statistical Analysis 3: Comparison: Part 2, Treatment D: Maribavir 200 mg vs Part 2, Treatment E: Rabeprazole 20 mg + Maribavir 200 mg; Comparison of AUClast of Maribavir: Part 2: Treatment E (Test) versus Treatment D (Reference); Test type: Other — A mixed-effects model was applied to ln-transformed plasma maribavir AUClast with treatment as a fixed effect, and participant as a random effect. Point estimates and their associated 90% CIs were constructed for the differences between Treatment E (test) versus Treatment D (reference). The point estimates and their associated 90% CIs were then back transformed to provide point estimates and 90% CIs for the ratios of Treatment E versus Treatment D; Geometric Mean Ratio (GMR) (%) = 70.00, 90% CI 2-sided [60.11 to 81.51] — GMR (%) was calculated as 100*(Test/Reference)

3. Primary Outcome: Parts 1 and 2: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity (AUC0-infinity) of Maribavir
Description: AUC0-infinity was defined as the area under the plasma concentration-time curve from time 0 to infinity of maribavir in plasma.
Time Frame: as for outcome 1
Population: PK set included all participants who received at least one dose of maribavir, did not vomit or had diarrhea within four hours of the maribavir dosing, and had five or more post-dose time points with evaluable post-dose maribavir concentration values that enabled NCA. Here, "Overall Number of Participants Analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg*h/mL
Arm/Group | Part 1, Treatment A: Maribavir 200 mg | Part 1, Treatment B: Maribavir 200 mg | Part 1, Treatment C: Maribavir 200 mg | Part 2, Treatment D: Maribavir 200 mg | Part 2, Treatment E: Rabeprazole 20 mg + Maribavir 200 mg
Number analyzed (Participants) | 18 | 18 | 18 | 14 | 10
mcg*h/mL | 59.1 (55.9) | 59.1 (56.3) | 48.2 (57.6) | 57.2 (38.5) | 50.1 (35.4)
Statistical Analysis 1: Comparison: Part 1, Treatment A: Maribavir 200 mg vs Part 1, Treatment B: Maribavir 200 mg; Comparison of AUC0-infinity of Maribavir: Part 1: Treatment B (Test) versus Treatment A (Reference); Test type: Other — A mixed-effects model was applied to ln-transformed plasma maribavir AUC0-infinity with treatment, period, and sequence as fixed effects, and participant within sequence as a random effect. Point estimates and their associated 90% CIs were constructed for differences between Treatment B (test) versus Treatment A (reference). Point estimates and their associated 90% CIs were then back transformed to provide point estimates and 90% CIs for ratios of Treatment B versus Treatment A; Geometric Mean Ratio (GMR) (%) = 99.94, 90% CI 2-sided [94.12 to 106.11] — GMR (%) was calculated as 100*(Test/Reference)
Statistical Analysis 2: Comparison: Part 1, Treatment B: Maribavir 200 mg vs Part 1, Treatment C: Maribavir 200 mg; Comparison of AUC0-infinity of Maribavir: Part 1: Treatment C (Test) versus Treatment B (Reference); Test type: Other — A mixed-effects model was applied to ln-transformed plasma maribavir AUC0-infinity with treatment, period, and sequence as fixed effects, and participant within sequence as a random effect. Point estimates and their associated 90% CIs were constructed for differences between Treatment C (test) versus Treatment B (reference). Point estimates and their associated 90% CIs were then back transformed to provide point estimates and 90% CIs for ratios of Treatment C versus Treatment B; Geometric Mean Ratio (GMR) (%) = 81.68, 90% CI 2-sided [76.93 to 86.73]
Statistical Analysis 3: Comparison: Part 2, Treatment D: Maribavir 200 mg vs Part 2, Treatment E: Rabeprazole 20 mg + Maribavir 200 mg; Comparison of AUC0-infinity of Maribavir: Part 2: Treatment E (Test) versus Treatment D (Reference); Test type: Other — A mixed-effects model was applied to ln-transformed plasma maribavir AUC0-infinity with treatment as a fixed effect, and participant as a random effect. Point estimates and their associated 90% CIs were constructed for the differences between Treatment E (test) versus Treatment D (reference). The point estimates and their associated 90% CIs were then back transformed to provide point estimates and 90% CIs for the ratios of Treatment E versus Treatment D; Geometric Mean Ratio (GMR) (%) = 88.92, 90% CI 2-sided [76.94 to 102.78] — GMR (%) was calculated as 100*(Test/Reference)

4. Secondary Outcome: Parts 1 and 2: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious TEAEs
Description: A TEAE was defined as an adverse event (AE) that was starting or worsening at the time of or after the first dose of maribavir administered in the study. An serious adverse event (SAE) was defined as any untoward medical occurrence that at any dose resulted in death; was life threatening; required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity; was a congenital anomaly/birth defect; was an important medical event that satisfies any of the following: might require intervention to prevent items 1 through 5 above and might exposed the participant to danger, even though the event is not immediately life threatening or fatal or does not result in hospitalization. Any clinically significant changes in vital signs, electrocardiogram (ECG) values and clinical laboratory parameters were considered as TEAEs.
Time Frame: Parts 1 and 2: From start of study drug administration up to follow-up (Day 16)
Population: Safety set included all participants who received at least one dose of maribavir.
Measure: Count of Participants; unit: Participants
Groups:
- Part 2, Treatment E1: Rabeprazole 20 mg: On Days 1 to 5 of Treatment Period 2, participants received oral doses of 20 mg rabeprazole, once daily, under fasting conditions.
- Part 2, Treatment E2: Maribavir 200 mg: On the morning of Day 5 of Treatment Period 2, two hours after rabeprazole dosing, participants received a single oral dose of 200 mg maribavir powder-for-oral suspension formulation under fasting conditions.
Arm/Group | Part 1, Treatment A: Maribavir 200 mg | Part 1, Treatment B: Maribavir 200 mg | Part 1, Treatment C: Maribavir 200 mg | Part 2, Treatment D: Maribavir 200 mg | Part 2, Treatment E1: Rabeprazole 20 mg | Part 2, Treatment E2: Maribavir 200 mg
Number analyzed (Participants) | 18 | 18 | 18 | 14 | 14 | 14
Participants
  TEAEs | 2 | 0 | 2 | 0 | 2 | 1
  Serious TEAEs | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Number of Participants Based on Severity of TEAEs
Description: Severity of TEAEs were determined by following criteria: Mild: An AE that was usually transient and might require only minimal treatment or therapeutic intervention. The event did not generally interfere with usual activities of daily living; Moderate: An AE that was usually alleviated with additional specific therapeutic intervention. The event interfered with usual activities of daily living, causing discomfort but possessed no significant or permanent risk of harm to the research participant; Severe: An AE that interrupted usual activities of daily living, or significantly affects clinical status, or might require intensive therapeutic intervention.
Time Frame: Parts 1 and 2: From start of study drug administration up to follow-up (Day 16)
Population: Safety set included all participants who received at least one dose of maribavir.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1, Treatment A: Maribavir 200 mg | Part 1, Treatment B: Maribavir 200 mg | Part 1, Treatment C: Maribavir 200 mg | Part 2, Treatment D: Maribavir 200 mg | Part 2, Treatment E1: Rabeprazole 20 mg | Part 2, Treatment E2: Maribavir 200 mg
Number analyzed (Participants) | 18 | 18 | 18 | 14 | 14 | 14
Participants
  Mild | 2 | 0 | 1 | 0 | 1 | 1
  Moderate | 0 | 0 | 1 | 0 | 1 | 0
  Severe | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Number of Participants Based on Causality of TEAEs
Description: The causality relationship of each AE to the study drug was assessed using the following categories: Related: An AE that followed a reasonable temporal sequence from administration of a drug (including the course after withdrawal of the drug), or for which a causal relationship was at least a reasonable possibility, that was, the relationship could not be ruled out, although factors other than the drug, such as underlying diseases, complications, concomitant drugs and concurrent treatments, might also be responsible; Not Related: An AE that did not follow a reasonable temporal sequence from administration of a drug and/or that could reasonably be explained by other factors, such as underlying diseases, complications, concomitant medications and concurrent treatments. Number of participants based on causality of TEAEs as assessed by the Investigator were reported.
Time Frame: Parts 1 and 2: From start of study drug administration up to follow-up (Day 16)
Population: Safety set included all participants who received at least one dose of maribavir.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1, Treatment A: Maribavir 200 mg | Part 1, Treatment B: Maribavir 200 mg | Part 1, Treatment C: Maribavir 200 mg | Part 2, Treatment D: Maribavir 200 mg | Part 2, Treatment E1: Rabeprazole 20 mg | Part 2, Treatment E2: Maribavir 200 mg
Number analyzed (Participants) | 18 | 18 | 18 | 14 | 14 | 14
Participants
  Related TEAEs | 1 | 0 | 1 | 0 | 0 | 0
  Not Related TEAEs | 1 | 0 | 1 | 0 | 2 | 1

ADVERSE EVENTS:
Time Frame: Parts 1 and 2: From start of study drug administration up to follow-up (Day 16)
Description: Safety set included all participants who received at least one dose of maribavir.
Arm/Group | Part 1, Treatment A: Maribavir 200 mg | Part 1, Treatment B: Maribavir 200 mg | Part 1, Treatment C: Maribavir 200 mg | Part 2, Treatment D: Maribavir 200 mg | Part 2, Treatment E1: Rabeprazole 20 mg | Part 2, Treatment E2: Maribavir 200 mg
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18 | 0/18 | 0/14 | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/18 | 0/14 | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 2/18 | 0/18 | 2/18 | 0/14 | 2/14 | 1/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1, Treatment A: Maribavir 200 mg (N=18) | Part 1, Treatment B: Maribavir 200 mg (N=18) | Part 1, Treatment C: Maribavir 200 mg (N=18) | Part 2, Treatment D: Maribavir 200 mg (N=14) | Part 2, Treatment E1: Rabeprazole 20 mg (N=14) | Part 2, Treatment E2: Maribavir 200 mg (N=14)
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Facial pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Urine odour abnormal (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-04-11): https://cdn.clinicaltrials.gov/large-docs/22/NCT05918822/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-06): https://cdn.clinicaltrials.gov/large-docs/22/NCT05918822/SAP_001.pdf